CLINICAL TRIAL: NCT04602000
Title: A Phase 2/3, Randomized, Parallel-group, Placebo-controlled, Double-Blind Study to Evaluate the Efficacy and Safety of CT-P59 in Combination With Standard of Care in Outpatients With SARS-CoV-2 Infection
Brief Title: A Phase 2/3 Study to Evaluate the Efficacy and Safety of CT-P59 in Patients With Mild to Moderate SARS-CoV-2 Infection
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Celltrion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CT-P59 3.2; 2020-003369-20 (EudraCT Number)
Record Dates: First submitted 2020-10-18; First posted 2020-10-26 (Actual); Results first posted 2022-07-20 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-06

CONDITIONS: SARS-CoV-2 Infection
MeSH Terms: conditions — COVID-19 | interventions — regdanvimab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- CT-P59 40 mg/kg group (Part 1) (Experimental): CT-P59 (regdanvimab), 40 mg/kg by IV infusion once
  Interventions: Biological: CT-P59
- CT-P59 80 mg/kg group (Part 1) (Experimental): CT-P59 (regdanvimab), 80 mg/kg by IV infusion once
  Interventions: Biological: CT-P59
- Placebo group (Part 1) (Placebo Comparator): Placebo, matching in volume of CT-P59 80 mg/kg by IV infusion once
  Interventions: Biological: Placebo
- CT-P59 40 mg/kg group (Part 2) (Experimental): CT-P59 (regdanvimab), 40 mg/kg by IV infusion once
  Interventions: Biological: CT-P59
- Placebo group (Part 2) (Placebo Comparator): Placebo, matching in volume of CT-P59 40 mg/kg by IV infusion once
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: CT-P59 — CT-P59 (40 mg/kg) by IV infusion administered over 90 minutes, once (Part 1)
  Other Names: regdanvimab
  Arms: CT-P59 40 mg/kg group (Part 1)
Biological: CT-P59 — CT-P59 (80 mg/kg) by IV infusion administered over 90 minutes, once (Part 1)
  Other Names: regdanvimab
  Arms: CT-P59 80 mg/kg group (Part 1)
Biological: Placebo — Placebo (80 mg/kg) by IV infusion administered over 90 minutes, once (Part 1)
  Arms: Placebo group (Part 1)
Biological: CT-P59 — CT-P59 (40 mg/kg) by IV infusion administered over 60 minutes, once (Part 2)
  Other Names: regdanvimab
  Arms: CT-P59 40 mg/kg group (Part 2)
Biological: Placebo — Placebo (40 mg/kg) by IV infusion administered over 60 minutes, once (Part 2)
  Arms: Placebo group (Part 2)

SUMMARY:
This was a Phase 2/3 study to assess the efficacy about therapeutic effect of CT-P59 to the mild to moderate SARS-CoV-2 infected patients and the safety during after study drug injection.

DETAILED DESCRIPTION:
CT-P59 is a human monoclonal antibody targeted against severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) spike protein as a treatment for SARS-CoV-2 infection, which is manufactured by recombinant deoxyribonucleic acid technology in a Chinese hamster ovary mammalian cell line. This Phase 2/3, randomized, parallel-group, placebo-controlled, double-blind study was designed to evaluate the safety, tolerability, and therapeutic potential of CT-P59 in outpatients with mild to moderate SARS-CoV-2 infection, not requiring supplemental oxygen therapy.

ELIGIBILITY:
Inclusion Criteria:

Patient had to meet all of the following criteria to be randomized in this study.

1. Patient was an adult male or female patient, aged 18 or above.
2. Patient was diagnosed with SARS-CoV-2 infection at Screening by using the sponsor-supplied rapid SARS-CoV-2 diagnostic test or RT-PCR (reverse transcription-polymerase chain reaction).
3. Patient with conditions meeting all of the following criteria:

   1. Oxygen saturation > 94% on room air.
   2. Not requiring supplemental oxygen.
4. Patient who had an onset of symptom no more than 7 days prior to the study drug administration.
5. Patient had 1 or more of the SARS-CoV-2 infection-associated symptoms within but no more than 7 days prior to the study drug administration.

Exclusion Criteria:

Patients meeting any of the following criteria were excluded from the study.

1. Patient had current severe condition meeting one of the following:

   1. Previous or current hospitalization or requirement of hospitalization for treatment of serious SARS-CoV-2 related conditions.
   2. Respiratory distress with respiratory rate ≥30 breaths/min.
   3. Required supplemental oxygen
   4. Experienced shock
   5. Complicated with other organs failure, and intensive care unit monitoring treatment is needed by investigator's discretion.
2. Patient had received or had a plan to receive any of the following prohibited medications or treatments:

   1. Drugs with actual or possible antiviral drugs and/or possible anti-SARS-CoV-2 activity including but not limited to remdesivir, chloroquine, hydroxychloroquine, dexamethasone (or alternative corticosteroids to dexamethasone), interferon beta-1b, ribavirin, and other immunomodulatory agents and human immunodeficiency virus protease inhibitors (lopinavir-ritonavir, etc.) for therapeutic purpose of SARS-CoV-2 infection prior to study drug administration
   2. Any SARS-CoV-2 human IV immunoglobulin, convalescent plasma for the treatment of SARS-CoV-2 infection prior to study drug administration
   3. Any other investigational device or medical product including but not limited to any monoclonal antibody (tocilizumab, sarilumab, etc.), fusion proteins or biologics for the treatment of SARS-CoV-2 infection prior to the study drug administration
   4. Use of medications that are contraindicated with SoC
   5. SARS-CoV-2 vaccine prior to the study drug administration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1642 (Actual)
Dates: Start 2020-10-05 (Actual); Primary Completion 2021-05-21 (Actual); Study Completion 2021-10-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Chungnam National University Hospital, Daejeon, Jung-gu, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kim JY, Sandulescu O, Preotescu LL, Rivera-Martinez NE, Dobryanska M, Birlutiu V, Miftode EG, Gaibu N, Caliman-Sturdza O, Florescu SA, Shi HJ, Streinu-Cercel A, Streinu-Cercel A, Lee SJ, Kim SH, Chang I, Bae YJ, Suh JH, Chung DR, Kim SJ, Kim MR, Lee SG, Park G, Eom JS. A Randomized Clinical Trial of Regdanvimab in High-Risk Patients With Mild-to-Moderate Coronavirus Disease 2019. Open Forum Infect Dis. 2022 Aug 8;9(8):ofac406. doi: 10.1093/ofid/ofac406. eCollection 2022 Aug. PMID 36043180
- [Derived] Hirsch C, Park YS, Piechotta V, Chai KL, Estcourt LJ, Monsef I, Salomon S, Wood EM, So-Osman C, McQuilten Z, Spinner CD, Malin JJ, Stegemann M, Skoetz N, Kreuzberger N. SARS-CoV-2-neutralising monoclonal antibodies to prevent COVID-19. Cochrane Database Syst Rev. 2022 Jun 17;6(6):CD014945. doi: 10.1002/14651858.CD014945.pub2. PMID 35713300
- [Derived] Streinu-Cercel A, Sandulescu O, Preotescu LL, Kim JY, Kim YS, Cheon S, Jang YR, Lee SJ, Kim SH, Chang I, Suh JH, Lee SG, Kim MR, Chung DR, Kim HN, Streinu-Cercel A, Eom JS. Efficacy and Safety of Regdanvimab (CT-P59): A Phase 2/3 Randomized, Double-Blind, Placebo-Controlled Trial in Outpatients With Mild-to-Moderate Coronavirus Disease 2019. Open Forum Infect Dis. 2022 Feb 2;9(4):ofac053. doi: 10.1093/ofid/ofac053. eCollection 2022 Apr. PMID 35295819
- [Derived] Kreuzberger N, Hirsch C, Chai KL, Tomlinson E, Khosravi Z, Popp M, Neidhardt M, Piechotta V, Salomon S, Valk SJ, Monsef I, Schmaderer C, Wood EM, So-Osman C, Roberts DJ, McQuilten Z, Estcourt LJ, Skoetz N. SARS-CoV-2-neutralising monoclonal antibodies for treatment of COVID-19. Cochrane Database Syst Rev. 2021 Sep 2;9(9):CD013825. doi: 10.1002/14651858.CD013825.pub2. PMID 34473343

RESULTS

PARTICIPANT FLOW:
Recruitment Details: For Part 1, participants were screened from 23 study centers in 4 countries and were enrolled from 23 study centers in 4 countries. For Part 2, participants were screened from 60 study centers in 14 countries and were enrolled from 58 study centers in 13 countries.
Pre-assignment Details: For Part 1, a total of 371 participants were screened and 327 participants were enrolled (44 screening failures) and randomized. For Part 2, a total of 1,467 participants were screened and 1,315 participants were enrolled (152 screening failures) and randomized.
Groups:
- CT-P59 40 mg/kg Group (Part 1); CT-P59 40 mg/kg Group (Part 2): Each participant received CT-P59 (regdanvimab) 40 mg/kg by IV infusion on Day 1.
- CT-P59 80 mg/kg Group (Part 1): Each participant received CT-P59 (regdanvimab) 80 mg/kg by IV infusion on Day 1.
- Placebo Group (Part 1): Each participant received placebo, matching in volume of CT-P59 80 mg/kg, by IV infusion on Day 1.
- Placebo Group (Part 2): Each participant received placebo, matching in volume of CT-P59 40 mg/kg, by IV infusion on Day 1.
Period: Overall Study
Arm/Group | CT-P59 40 mg/kg Group (Part 1) | CT-P59 80 mg/kg Group (Part 1) | Placebo Group (Part 1) | CT-P59 40 mg/kg Group (Part 2) | Placebo Group (Part 2)
Started | 105 | 111 | 111 | 656 | 659
Completed | 97 | 103 | 105 | 618 | 608
Not Completed | 8 | 8 | 6 | 38 | 51
Not completed — Withdrawal by Subject | 3 | 6 | 3 | 27 | 39
Not completed — Physician Decision | 1 | 0 | 0 | 2 | 2
Not completed — Death | 0 | 1 | 0 | 1 | 2
Not completed — Lost to Follow-up | 0 | 0 | 0 | 3 | 4
Not completed — Other | 4 | 1 | 2 | 5 | 4
Not completed — Completed Treatment Period but not entered into Follow-up Period | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CT-P59 40 mg/kg Group (Part 1) | CT-P59 80 mg/kg Group (Part 1) | Placebo Group (Part 1) | CT-P59 40 mg/kg Group (Part 2) | Placebo Group (Part 2) | Total
Number analyzed (Participants) | 105 | 111 | 111 | 656 | 659 | 1642
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 0 | 0 | 1 | 5 | 7
  Between 18 and 65 years | 89 | 90 | 93 | 562 | 576 | 1410
  >=65 years | 15 | 21 | 18 | 93 | 78 | 225
Age, Continuous [Median (Full Range); unit: years] | 51.0 [18 to 75] | 51.0 [23 to 85] | 52.0 [23 to 88] | 49.0 [18 to 87] | 47.0 [18 to 83] | 49.0 [18 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46 | 52 | 63 | 309 | 332 | 802
  Male | 59 | 59 | 48 | 347 | 327 | 840
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 94 | 96 | 96 | 563 | 569 | 1418
  African American/Black | 0 | 0 | 0 | 6 | 1 | 7
  American Indian/Alaska native | 0 | 0 | 0 | 5 | 9 | 14
  Asian | 11 | 15 | 15 | 7 | 7 | 55
  Native Hawaiian/Other Pacific Islander | 0 | 0 | 0 | 1 | 0 | 1
  Not allowed by investigator country regulations | 0 | 0 | 0 | 0 | 0 | 0
  Other | 0 | 0 | 0 | 74 | 73 | 147
Region of Enrollment [Number; unit: participants]
  Hungary | 0 | 0 | 0 | 25 | 32 | 57
  Italy | 0 | 0 | 0 | 2 | 2 | 4
  South Korea | 11 | 15 | 14 | 6 | 6 | 52
  North Macedonia | 0 | 0 | 0 | 30 | 26 | 56
  Mexico | 0 | 0 | 0 | 68 | 70 | 138
  Moldova | 0 | 0 | 0 | 19 | 18 | 37
  Peru | 0 | 0 | 0 | 11 | 9 | 20
  Poland | 0 | 0 | 0 | 43 | 47 | 90
  Romania | 93 | 90 | 93 | 315 | 311 | 902
  Serbia | 0 | 0 | 0 | 23 | 24 | 47
  Spain | 0 | 2 | 1 | 7 | 14 | 24
  Ukraine | 0 | 0 | 0 | 58 | 49 | 107
  United States | 1 | 4 | 3 | 49 | 51 | 108

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients With Clinical Symptom Requiring Hospitalization, Oxygen Therapy, or Experiencing Mortality Due to SARS-CoV-2 Infection (Part 1)
Description: To assess the clinically meaningful therapeutic efficacy of CT-P59 as determined by proportion of patients with clinical symptom requiring hospitalization, oxygen therapy, or experiencing mortality due to SARS-CoV-2 infection up to Day 28
Time Frame: Up to Day 28
Population: ITTI Set (defined as all randomly assigned patients with confirmed SARS-CoV-2 infection by pre-infusion result [Day 1] of RT-qPCR and who received a complete or partial dose of the study drug; Patient who had confirmed negative or missing at Day 1 and positive at Day 2 was also included)
Measure: Count of Participants; unit: Participants
Arm/Group | CT-P59 40 mg/kg Group (Part 1) | CT-P59 80 mg/kg Group (Part 1) | Placebo Group (Part 1)
Number analyzed (Participants) | 101 | 103 | 103
Participants | 4 | 5 | 9

2. Primary Outcome: Proportion of Patients With Negative Conversion in Nasopharyngeal Swab Specimen Based on RT-qPCR at Each Visit (Part 1)
Description: To assess the potential therapeutic efficacy of CT-P59 as determined by proportion of negative conversion in nasopharyngeal swab specimen based on RT-qPCR up to Day 14
Time Frame: Up to Day 14
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | CT-P59 40 mg/kg Group (Part 1) | CT-P59 80 mg/kg Group (Part 1) | Placebo Group (Part 1)
Number analyzed (Participants) | 101 | 103 | 103
Participants
  Day 2 | 0 | 1 | 0
  Day 3 | 4 | 4 | 3
  Day 4 | 2 | 6 | 4
  Day 5 | 7 | 3 | 2
  Day 6 | 5 | 5 | 4
  Day 7 | 8 | 12 | 7
  Day 10 | 19 | 18 | 19
  Day 14 | 23 | 19 | 23

3. Primary Outcome: Time to Negative Conversion in Nasopharyngeal Swab Specimen (Part 1)
Description: To evaluate the therapeutic efficacy of CT-P59 as determined by time to negative conversion by RT-qPCR up to Day 14
Time Frame: Up to Day 14
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | CT-P59 40 mg/kg Group (Part 1) | CT-P59 80 mg/kg Group (Part 1) | Placebo Group (Part 1)
Number analyzed (Participants) | 101 | 103 | 103
days | 12.75 [9.00 to 12.84] | 11.89 [8.94 to 12.91] | 12.94 [12.75 to 13.99]

4. Primary Outcome: Time to Clinical Recovery (Part 1)
Description: To assess the potential therapeutic efficacy of CT-P59 as determined by time to clinical recovery up to Day 14.
  Clinical recovery was defined as all symptoms on the SARS-CoV-2 Infection Symptom Checklist 1 being recorded as 'absent' or 'mild' in intensity for at least 48 hours. SARS-CoV-2 Infection Symptom Checklist 1 consisted of 7 symptoms (feeling feverish, cough, shortness of breath or difficulty breathing, sore throat, body pain or muscle pain, fatigue, and headache) and the intensity of patient's self-aware for each SARS-CoV-2 infection symptom (absent [0], mild [1]. moderate [2], and severe [3]).
  To meet the clinical recovery, symptoms 'severe' or 'moderate' in intensity at baseline should be changed to 'mild' or 'absent', or symptoms 'mild' in intensity at baseline should be changed to 'absent', after the study drug administration. Symptoms "absent" in intensity at baseline should maintain as "absent" for at least 48 hours.
Time Frame: Up to Day 14
Population: ITTI Set (defined as all randomly assigned patients with confirmed SARS-CoV-2 infection by pre-infusion result [Day 1] of RT-qPCR and who received a complete or partial dose of the study drug; Patient who had confirmed negative or missing at Day 1 and positive at Day 2 was also included; Patients who have absent for all symptoms or at least one missing at baseline are excluded.)
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | CT-P59 40 mg/kg Group (Part 1) | CT-P59 80 mg/kg Group (Part 1) | Placebo Group (Part 1)
Number analyzed (Participants) | 95 | 92 | 98
days | 7.18 [5.50 to 9.37] | 7.30 [5.72 to 9.33] | 8.80 [6.88 to 13.09]

5. Primary Outcome: Proportion of Patients With Clinical Symptom Requiring Hospitalization, Oxygen Therapy, or Experiencing Mortality Due to SARS-CoV-2 Infection up to Day 28 in High-risk Patients (Part 2)
Description: To demonstrate the clinically meaningful therapeutic efficacy of CT-P59 as determined by proportion of patients with clinical symptom requiring hospitalization, oxygen therapy, or experiencing mortality due to SARS-CoV-2 infection up to Day 28 in high-risk patients
Time Frame: Up to Day 28
Population: ITT Set - High Risk (defined as all randomly assigned patients to the study drug, who were at high-risk for progressing to severe COVID-19 and/or hospitalization and who met at least 1 of the high-risk criteria)
Measure: Count of Participants; unit: Participants
Arm/Group | CT-P59 40 mg/kg Group (Part 2) | Placebo Group (Part 2)
Number analyzed (Participants) | 446 | 434
Participants | 14 | 48
Statistical Analysis 1: Comparison: CT-P59 40 mg/kg Group (Part 2) vs Placebo Group (Part 2); Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; P-value was calculated using CMH test stratified by age (≥60 vs. <60 years), baseline comorbidities (Yes vs. No) and region (US vs. EU vs. Other); Difference estimated using CMH weights = -8.0, 95% CI 2-sided [-11.7 to -4.5] — The 95% stratified Newcombe CI with CMH weights was presented

6. Secondary Outcome: Proportion of Patients With Clinical Symptom Requiring Hospitalization, Oxygen Therapy, or Experiencing Mortality Due to SARS-CoV-2 Infection up to Day 28 in All Randomized Patients (Part 2)
Description: To demonstrate the clinically meaningful therapeutic efficacy of CT-P59 as determined by proportion of patients with clinical symptom requiring hospitalization, oxygen therapy, or experiencing mortality due to SARS-CoV-2 infection up to Day 28 in all randomized patients
Time Frame: Up to Day 28
Population: ITT Set (defined as all randomly assigned patients to the study drug)
Measure: Count of Participants; unit: Participants
Arm/Group | CT-P59 40 mg/kg Group (Part 2) | Placebo Group (Part 2)
Number analyzed (Participants) | 656 | 659
Participants | 16 | 53

7. Secondary Outcome: Time to Clinical Recovery up to Day 14 in High-risk Patients (Part 2)
Description: To assess the potential therapeutic efficacy of CT-P59 as determined by time to clinical recovery up to Day 14 in high-risk patients.
  Clinical recovery was defined as all symptoms on the SARS-CoV-2 Infection Symptom Checklist 1 being recorded as 'absent' or 'mild' in intensity for at least 48 hours. SARS-CoV-2 Infection Symptom Checklist 1 consisted of 7 symptoms (feeling feverish, cough, shortness of breath or difficulty breathing, sore throat, body pain or muscle pain, fatigue, and headache) and the intensity of patient's self-aware for each SARS-CoV-2 infection symptom (absent [0], mild [1]. moderate [2], and severe [3]).
  To meet the clinical recovery, symptoms 'severe' or 'moderate' in intensity at baseline should be changed to 'mild' or 'absent', or symptoms 'mild' in intensity at baseline should be changed to 'absent', after the study drug administration. Symptoms "absent" in intensity at baseline should maintain as "absent" for at least 48 hours.
Time Frame: Up to Day 14
Population: ITT Set - High Risk (defined as all randomly assigned patients to the study drug, who were at high-risk for progressing to severe COVID-19 and/or hospitalization and who met at least 1 of the high-risk criteria; Patient who reported at least 1 symptom at baseline was included)
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | CT-P59 40 mg/kg Group (Part 2) | Placebo Group (Part 2)
Number analyzed (Participants) | 429 | 406
days | 9.27 [8.27 to 11.05] | NA [12.35 to NA] — The median time in Placebo group was not reached as less than 50% of patients achieved clinical recovery and the number of patients achieved clinical recovery in Placebo group was not sufficient to calculate the upper CI.

8. Secondary Outcome: Time to Clinical Recovery up to Day 14 in All Randomized Patients (Part 2)
Description: To assess the potential therapeutic efficacy of CT-P59 as determined by time to clinical recovery up to Day 14 in all randomized patients.
  Clinical recovery was defined as all symptoms on the SARS-CoV-2 Infection Symptom Checklist 1 being recorded as 'absent' or 'mild' in intensity for at least 48 hours. SARS-CoV-2 Infection Symptom Checklist 1 consisted of 7 symptoms (feeling feverish, cough, shortness of breath or difficulty breathing, sore throat, body pain or muscle pain, fatigue, and headache) and the intensity of patient's self-aware for each SARS-CoV-2 infection symptom (absent [0], mild [1]. moderate [2], and severe [3]).
  To meet the clinical recovery, symptoms 'severe' or 'moderate' in intensity at baseline should be changed to 'mild' or 'absent', or symptoms 'mild' in intensity at baseline should be changed to 'absent', after the study drug administration. Symptoms "absent" in intensity at baseline should maintain as "absent" for at least 48 hours.
Time Frame: Up to Day 14
Population: ITT Set (defined as all randomly assigned patients to the study drug; Patient who reported at least 1 symptom at baseline was included)
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | CT-P59 40 mg/kg Group (Part 2) | Placebo Group (Part 2)
Number analyzed (Participants) | 629 | 618
days | 8.38 [7.91 to 9.33] | 13.25 [11.94 to NA] — The number of patients achieved clinical recovery in Placebo group was not sufficient to calculate the upper CI.

9. Secondary Outcome: Proportion of Patients With Hospital Admission Due to SARS-CoV-2 Infection (Part 1 and Part 2)
Description: To evaluate the additional efficacy of CT-P59
Time Frame: Up to Day 28
Population: ITTI Set for Part 1 (defined as all randomly assigned patients with confirmed SARS-CoV-2 infection by pre-infusion result [Day 1] of RT-qPCR and who received a complete or partial dose of the study drug; Patient who had confirmed negative or missing at Day 1 and positive at Day 2 was also included) and ITT Set for Part 2 (defined as all randomly assigned patients to study drug)
Measure: Count of Participants; unit: Participants
Arm/Group | CT-P59 40 mg/kg Group (Part 1) | CT-P59 80 mg/kg Group (Part 1) | Placebo Group (Part 1) | CT-P59 40 mg/kg Group (Part 2) | Placebo Group (Part 2)
Number analyzed (Participants) | 101 | 103 | 103 | 656 | 659
Participants | 4 | 5 | 9 | 16 | 52

10. Secondary Outcome: Proportion of Patients Requiring Supplemental Oxygen Due to SARS-CoV-2 Infection (Part 1 and Part 2)
Description: To evaluate the additional efficacy of CT-P59
Time Frame: Up to Day 28
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | CT-P59 40 mg/kg Group (Part 1) | CT-P59 80 mg/kg Group (Part 1) | Placebo Group (Part 1) | CT-P59 40 mg/kg Group (Part 2) | Placebo Group (Part 2)
Number analyzed (Participants) | 101 | 103 | 103 | 656 | 659
Participants | 4 | 4 | 9 | 15 | 49

11. Secondary Outcome: Proportion of Patients With Mechanical Ventilation Use Due to SARS-CoV-2 Infection (Part 1 and Part 2)
Description: To evaluate the additional efficacy of CT-P59
Time Frame: Up to Day 28
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | CT-P59 40 mg/kg Group (Part 1) | CT-P59 80 mg/kg Group (Part 1) | Placebo Group (Part 1) | CT-P59 40 mg/kg Group (Part 2) | Placebo Group (Part 2)
Number analyzed (Participants) | 101 | 103 | 103 | 656 | 659
Participants | 0 | 1 | 0 | 0 | 3

12. Secondary Outcome: Proportion of Patients Requiring Rescue Therapy Due to SARS-CoV-2 Infection (Part 1 and Part 2)
Description: To evaluate the additional efficacy of CT-P59
Time Frame: Up to Day 28
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | CT-P59 40 mg/kg Group (Part 1) | CT-P59 80 mg/kg Group (Part 1) | Placebo Group (Part 1) | CT-P59 40 mg/kg Group (Part 2) | Placebo Group (Part 2)
Number analyzed (Participants) | 101 | 103 | 103 | 656 | 659
Participants | 7 | 11 | 15 | 37 | 85

13. Secondary Outcome: Proportion of Patients With Intensive Care Unit Transfer Due to SARS-CoV-2 Infection (Part 1 and Part 2)
Description: To evaluate the additional efficacy of CT-P59
Time Frame: Up to Day 28
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | CT-P59 40 mg/kg Group (Part 1) | CT-P59 80 mg/kg Group (Part 1) | Placebo Group (Part 1) | CT-P59 40 mg/kg Group (Part 2) | Placebo Group (Part 2)
Number analyzed (Participants) | 101 | 103 | 103 | 656 | 659
Participants | 0 | 0 | 0 | 0 | 5

14. Secondary Outcome: Proportion of Patients With All-cause Mortality (Part 1 and Part 2)
Description: To evaluate the additional efficacy of CT-P59
Time Frame: Up to Day 28
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | CT-P59 40 mg/kg Group (Part 1) | CT-P59 80 mg/kg Group (Part 1) | Placebo Group (Part 1) | CT-P59 40 mg/kg Group (Part 2) | Placebo Group (Part 2)
Number analyzed (Participants) | 101 | 103 | 103 | 656 | 659
Participants | 0 | 0 | 0 | 1 | 2

15. Secondary Outcome: Time to Negative Conversion in Nasopharyngeal Swab Specimen Based on RT-qPCR (Part 1 and Part 2)
Description: To evaluate the additional efficacy of CT-P59
Time Frame: Up to Day 28
Population: ITTI Set for Part 1 (defined as all randomly assigned patients with confirmed SARS-CoV-2 infection by pre-infusion result [Day 1] of RT-qPCR and who received a complete or partial dose of the study drug; Patient who had confirmed negative or missing at Day 1 and positive at Day 2 was also included) and ITT Set for Part 2 (defined as all randomly assigned patients to study drug; Patient who had positive result confirmed based on the negative threshold at baseline was included)
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | CT-P59 40 mg/kg Group (Part 1) | CT-P59 80 mg/kg Group (Part 1) | Placebo Group (Part 1) | CT-P59 40 mg/kg Group (Part 2) | Placebo Group (Part 2)
Number analyzed (Participants) | 101 | 103 | 103 | 612 | 618
days | 12.75 [9.00 to 12.84] | 11.89 [8.94 to 12.91] | 12.94 [12.75 to 13.99] | 11.90 [9.02 to 12.83] | 13.15 [12.97 to 18.80]

16. Secondary Outcome: Proportion of Patient With Negative Conversion in Nasopharyngeal Swab Specimen Based on RT-qPCR at Each Visit (Part 1 and Part 2)
Description: To evaluate the additional efficacy of CT-P59
Time Frame: Days 3, 7, 10, 14, 21, and 28
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | CT-P59 40 mg/kg Group (Part 1) | CT-P59 80 mg/kg Group (Part 1) | Placebo Group (Part 1) | CT-P59 40 mg/kg Group (Part 2) | Placebo Group (Part 2)
Number analyzed (Participants) | 101 | 103 | 103 | 612 | 618
Participants
  Day 3 | 4 | 4 | 3 | 34 | 21
  Day 7 | 8 | 12 | 7 | 141 | 94
  Day 10 | 19 | 18 | 19 | 137 | 117
  Day 14 | 23 | 19 | 23 | 113 | 149
  Day 21 | 10 | 8 | 9 | 99 | 117
  Day 28 | 6 | 5 | 5 | 52 | 61

17. Secondary Outcome: Time to Clinical Recovery (Part 1 and Part 2)
Description: To evaluate the additional efficacy of CT-P59. Clinical recovery was defined as all symptoms on the SARS-CoV-2 Infection Symptom Checklist 1 being recorded as 'absent' or 'mild' in intensity for at least 48 hours. SARS-CoV-2 Infection Symptom Checklist 1 consisted of 7 symptoms (feeling feverish, cough, shortness of breath or difficulty breathing, sore throat, body pain or muscle pain, fatigue, and headache) and the intensity of patient's self-aware for each SARS-CoV-2 infection symptom (absent [0], mild [1]. moderate [2], and severe [3]).
  To meet the clinical recovery, symptoms 'severe' or 'moderate' in intensity at baseline should be changed to 'mild' or 'absent', or symptoms 'mild' in intensity at baseline should be changed to 'absent', after the study drug administration. Symptoms "absent" in intensity at baseline should maintain as "absent" for at least 48 hours.
Time Frame: Up to Day 28
Population: ITTI Set for Part 1 (all randomly assigned patients with confirmed SARS-CoV-2 infection by Day 1 of RT-qPCR and who received a complete or partial dose of the study drug; Patient who had confirmed negative or missing at Day 1 and positive at Day 2 was also included; Patients who had absent for all symptoms or at least one missing at baseline are excluded), and ITT Set for Part 2 (all randomly assigned patients to study drug; Patient who reported at least 1 symptom at baseline was included)
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | CT-P59 40 mg/kg Group (Part 1) | CT-P59 80 mg/kg Group (Part 1) | Placebo Group (Part 1) | CT-P59 40 mg/kg Group (Part 2) | Placebo Group (Part 2)
Number analyzed (Participants) | 95 | 92 | 98 | 629 | 618
days | 7.18 [5.50 to 9.37] | 7.30 [5.72 to 9.33] | 8.80 [6.88 to 13.09] | 8.39 [8.01 to 9.39] | 13.29 [12.12 to 15.25]

18. Other Pre Specified Outcome: [Virology] Viral Serology for SARS-CoV-2 Antibody
Description: To assess the serology of SARS-CoV-2 antibody. The proportions of patients positive with IgG or IgM were summarized.
Time Frame: Days 1, 7, 14, 28, and 56
Population: ITTI Set (defined as all randomly assigned patients with confirmed SARS-CoV-2 infection by pre-infusion result (Day 1) of RT-qPCR, who receive a complete or partial dose of study drug) for both Parts.
Measure: Count of Participants; unit: Participants
Arm/Group | CT-P59 40 mg/kg Group (Part 1) | CT-P59 80 mg/kg Group (Part 1) | Placebo Group (Part 1) | CT-P59 40 mg/kg Group (Part 2) | Placebo Group (Part 2)
Number analyzed (Participants) | 101 | 103 | 103 | 612 | 618
Participants
  IgG - Day 1 | 0 | 6 | 3 | 45 | 35
  IgG - Day 7 | 27 | 32 | 32 | 354 | 322
  IgG - Day 14 | 77 | 82 | 86 | 498 | 509
  IgG - Day 28 | 84 | 94 | 91 | 535 | 548
  IgG - Day 56 | 78 | 85 | 86 | 506 | 532
  IgM - Day 1 | 2 | 6 | 4 | 53 | 55
  IgM - Day 7 | 38 | 43 | 49 | 362 | 332
  IgM - Day 14 | 78 | 82 | 87 | 467 | 491
  IgM - Day 28 | 59 | 77 | 65 | 461 | 493
  IgM - Day 56 | 39 | 54 | 51 | 407 | 441

19. Other Pre Specified Outcome: [PK] Area Under the Concentration-time Curve From Time Zero to Infinity (AUC0-inf) (Part 1)
Description: To assess the PK of CT-P59
Time Frame: Pre-dose, end of infusion, 1, 24, 48, 96, 144, 216, 312, 648, 1320, 2136 hours after start of infusion
Population: PK Set (defined as all randomly assigned patients with confirmed SARS-CoV-2 infection by pre-infusion [Day 1] result based on RT-qPCR and who had signed informed consent to participate in a PK sub-study, received a complete dose of study drug, and had at least 1 evaluable post-treatment PK result; If the pre-infusion result at Day 1 was confirmed negative or missing and the Day 2 result was confirmed positive, this patient was also included)
Measure: Mean (Standard Deviation); unit: h*μg/mL
Arm/Group | CT-P59 40 mg/kg Group (Part 1) | CT-P59 80 mg/kg Group (Part 1)
Number analyzed (Participants) | 29 | 32
h*μg/mL | 212460.507 (46724.5556) | 426694.643 (121171.182)

20. Other Pre Specified Outcome: [PK] Maximum Serum Concentration (Cmax) (Part 1)
Description: To assess the PK of CT-P59
Time Frame: Pre-dose, end of infusion, 1, 24, 48, 96, 144, 216, 312, 648, 1320, 2136 hours after start of infusion
Population: PK Set (defined as all randomly assigned patients with confirmed SARS-CoV-2 infection by pre-infusion (Day 1) result based on RT-qPCR and who had signed informed consent to participate in a PK sub-study, received a complete dose of study drug, and had at least 1 evaluable post-treatment PK result)
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | CT-P59 40 mg/kg Group (Part 1) | CT-P59 80 mg/kg Group (Part 1)
Number analyzed (Participants) | 29 | 32
μg/mL | 1016.6 (268.97) | 2007.6 (477.97)

21. Other Pre Specified Outcome: [PK] Terminal Half-life (t1/2) (Part 1)
Description: To assess the PK of CT-P59
Time Frame: Pre-dose, end of infusion, 1, 24, 48, 96, 144, 216, 312, 648, 1320, 2136 hours after start of infusion
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: h
Arm/Group | CT-P59 40 mg/kg Group (Part 1) | CT-P59 80 mg/kg Group (Part 1)
Number analyzed (Participants) | 29 | 32
h | 403.916 (147.8450) | 453.442 (107.5620)

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) and serious adverse events (SAEs) were reported by the investigator from the date patients signed the informed consent form (ICF) until the last assessment date or End-of-Treatment (EOT) visit (Period: day of ICF signed to Day 90[EOT]), regardless of the relationship to the study drug.
Description: The investigator was responsible for reporting all AEs that were observed or reported from signing of ICF to EOT, regardless of their relationship to study drug or their clinical significance.
  Cases of worsening of SARS-CoV-2 infection which were considered as unrelated to the study drug were not collected and not reported as an (S)AE.
  The analysis population is Safety Set and it is defined as all randomly assigned patients who received a complete or partial dose of the study drug.
  All-cause
Arm/Group | CT-P59 40 mg/kg Group (Part 1) | CT-P59 80 mg/kg Group (Part 1) | Placebo Group (Part 1) | CT-P59 40 mg/kg Group (Part 2) | Placebo Group (Part 2)
All-Cause Mortality (participants affected / at risk) | 0/105 | 0/110 | 0/110 | 1/652 | 2/650
Serious Adverse Events (participants affected / at risk) | 0/105 | 0/110 | 0/110 | 6/652 | 5/650
Other Adverse Events (participants affected / at risk) | 19/105 | 18/110 | 17/110 | 119/652 | 128/650
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CT-P59 40 mg/kg Group (Part 1) (N=105) | CT-P59 80 mg/kg Group (Part 1) (N=110) | Placebo Group (Part 1) (N=110) | CT-P59 40 mg/kg Group (Part 2) (N=652) | Placebo Group (Part 2) (N=650)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Angina unstable (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hiatus hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intraocular melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CT-P59 40 mg/kg Group (Part 1) (N=105) | CT-P59 80 mg/kg Group (Part 1) (N=110) | Placebo Group (Part 1) (N=110) | CT-P59 40 mg/kg Group (Part 2) (N=652) | Placebo Group (Part 2) (N=650)
Leukopenia (Blood and lymphatic system disorders) | 3 (3) | 3 (3) | 0 (0) | 6 (6) | 12 (12)
Thrombocytosis (Blood and lymphatic system disorders) | 3 (3) | 1 (1) | 2 (2) | 11 (11) | 5 (5)
Cystitis (Infections and infestations) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (2) | 1 (1) | 19 (22) | 31 (34)
Blood creatine phosphokinase increased (Investigations) | 5 (5) | 2 (2) | 1 (1) | 14 (14) | 10 (10)
C-reactive protein increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 18 (18) | 10 (10)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 1 (1) | 1 (2) | 8 (8) | 20 (20)
Hepatic enzyme increased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 21 (21) | 15 (16)
Inflammatory marker increased (Investigations) | 0 (0) | 3 (3) | 2 (2) | 14 (14) | 17 (18)
Dyslipidaemia (Metabolism and nutrition disorders) | 4 (4) | 3 (3) | 2 (2) | 7 (7) | 9 (9)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2) | 3 (4) | 12 (12) | 9 (9)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 3 (5) | 2 (2) | 9 (10) | 6 (7)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 6 (7) | 0 (0) | 3 (5) | 29 (35) | 33 (40)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 2 (2)
Insomnia (Psychiatric disorders) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 5 (5)
Hypertension (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 17 (22) | 14 (15)
Bacteriuria (Infections and infestations) | 2 (2) | 2 (2) | 2 (2) | 3 (3) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (3):
  • Study Protocol (2021-04-30): https://cdn.clinicaltrials.gov/large-docs/00/NCT04602000/Prot_003.pdf
  • Statistical Analysis Plan: Part 1 (2021-07-22): https://cdn.clinicaltrials.gov/large-docs/00/NCT04602000/SAP_004.pdf
  • Statistical Analysis Plan: Part 2 (2021-12-16): https://cdn.clinicaltrials.gov/large-docs/00/NCT04602000/SAP_005.pdf